CLINICAL TRIAL: NCT02855814
Title: Body Composition Reference Data for Preterm Infants
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: Santa Clara Valley Medical Center (Other); Baystate Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 1001M76732
Record Dates: First submitted 2016-07-27; First posted 2016-08-04 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth | interventions — Body Composition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Body Composition — No intervention. This is an observational, normative study of body composition variation in preterm infants

SUMMARY:
The American Academy of Pediatrics has recommended that growth in size (weight, length, and head circumference) and in body composition (fat and lean mass) in preterm infants should adhere as close as possible to the growth and body composition of a healthy infant in utero at the same gestational age. However, there are no body composition reference curves available at this time for the preterm infant population. The purpose of this study is to collect cross-sectional body composition data using air displacement plethysmography (PEA POD Infant Body Composition System, Life Measurement, Inc) on approximately 240 preterm infants within 3 days of birth, for the purpose of generating means, standard deviations, and percentile values for total body fat mass, total fat free mass, and percent body fat for infants born at 30-36 weeks gestation. Relatively healthy infants without evidence of growth retardation will be selected for form the reference sample. The goal is to generate a set of common reference curves to be used in clinical centers against which to compare body composition status for individual infants.

ELIGIBILITY:
Inclusion Criteria:

* Appropriate for gestational age (AGA), singleton, 30+0 and 36+6 weeks gestational age

Exclusion Criteria:

* Congenital defects that affect growth
* Inability to tolerate room air for 5 minutes without desaturation or bradycardia
* <1 kg birth weight
* Parents did not provide consent

Ages: 24 Hours to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: AGA, singleton, healthy infants born between 30+0 and 36+6 weeks gestation were eligible. The study was conducted between 2010 and 2015 at three tertiary NICU's in the United States: the University of Minnesota Masonic Children's Hospital in Minneapolis, MN (referred to hereafter as the MN site), Santa Clara Valley Medical Center in San Jose, CA (referred to as the SC site), and Baystate Medical Center in Springfield, MA (referred to as BS).
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Fat mass | Within 72 hours of birth
  Total body fat mass measured by air displacement plethysmography, in kg
Fat-free mass | Within 72 hours of birth
  Total body fat-free mass measured by air displacement plethysmography, in kg
Percent body fat | Within 72 hours of birth
  Percent body fat measured by air displacement plethysmography, in %

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Demerath EW, Johnson W, Davern BA, Anderson CG, Shenberger JS, Misra S, Ramel SE. New body composition reference charts for preterm infants. Am J Clin Nutr. 2017 Jan;105(1):70-77. doi: 10.3945/ajcn.116.138248. Epub 2016 Nov 2. PMID 27806978